CLINICAL TRIAL: NCT04170777
Title: Use of Cone-beam Computed Tomography on Gamma Knife Perfexion for Stereotactic Radiosurgery
Brief Title: Perfexion Registration Using CBCT
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 17-5662
Record Dates: First submitted 2019-11-12; First posted 2019-11-20 (Actual); Last update posted 2023-01-26 (Actual); Status verified 2023-01

CONDITIONS: Brain Metastases
Keywords: Advanced cancer; Imaging study; Stereotactic Radiosurgery; GammaKnife; Cone-beam computed tomography (CBCT)
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: The CBCT imaging involved for Arm A is considered part of the study treatment. Pre and post treatment images will be acquired of the patient treated on Perfexion Gamma Knife using the 'Leksell Coordinate Frame'.
- Arm B: Arm B will be undergoing standard treatment on Gamma Knife Perfexion for Stereotactic Radiosurgery using the 'relocatable mask'. Patients with lesions that are >3 cm at the largest diameter will be treated with the relocatable mask for which a hypo fractionated approach may be beneficial.

SUMMARY:
Measuring precision radiation delivery through cone-beam computed tomography (CBCT) and intra-fraction motion management (IFMM) incorporated on a GammaKnife unit via the Leksell Coordinate Frame (LCF) and relocatable mask system (RMS) immobilization devices.

DETAILED DESCRIPTION:
: Brain metastases are reported to occur in 20% to 40% of all patients with cancer. Treatment options for brain metastases include surgical resection, particularly in lesions causing significant mass effect, whole brain radiation (WBRT) and radiosurgery (SRS). Due to concerns of neurocognitive toxicity following WBRT, there is growing use of SRS, particularly in patients with limited brain metastases and controlled extracranial disease.

Radiosurgery delivers a high dose of radiation to a defined intracranial target through precise targeting with a sharp dose fall off at the target boundaries and minimal damage to surrounding tissue. To date, precision radiation delivery has been facilitated through the Leksell Coordinate Frame (LCF), fixated to the patient's skull through 4 pins. A relocatable mask system (RMS), consisting of a patient specific head rest and mask was developed to enable minimally-invasive fractioned radiosurgery.

A cone-beam computed tomography (CBCT) image guidance and intra-fraction motion management (IFMM) system was previously developed in-house in order to measure and address setup uncertainties on Gamma Knife. The in-house prototype has been integrated into a commercially available GammaKnife device with CBCT guidance. The installation of this device will enable volumetric guidance for all patients treated in either a single or multiple session on GammaKnife Perfexion.

This study is designed to have 2 arms, A and B. Both Arm A (using the Leksell Coordinate Frame) and Arm B (using the relocatable mask) are undergoing standard of care treatment on GammaKnife Perfexion for SRS. CBCT is part of standard of care for Arm B. However, CBCT imaging is considered as part of study treatment for Arm A. Pre and post treatment images will be acquired of the patient treated on Perfexion Gamma Knife using the Leksell Coordinate Frame in order to aid in analyzing the imaging metrics of the Image Guided Perfexion unit.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years old
2. Ability to provide informed consent
3. Any patient receiving single or multi-fraction stereotactic radiosurgery on the Perfexion Gamma Knife with image-guidance

Exclusion Criteria:

1. Age < 18 years old.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Brain metastases scheduled to receive SRS treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1250 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2022-09-29 (Actual)

PRIMARY OUTCOMES:
Setup variation of LCF and relocatable mask using CBCT Imaging | Through study completion, an average of 1 week
  To quantify inter- and intra-fraction setup variations with the Leksell Coordinate Frame (LCF) and relocatable mask device as measured on CBCT and IFMM
Setup variation in positioning between CT planning and treatment | Through study completion, an average of 1 week
  Measure intra-fraction setup variations between the CT planning and treatment position for the LCF and relocatable mask device

SECONDARY OUTCOMES:
Target volume margins for brain metastases | Through study completion, an average of 1 week
  To determine evidence-based planning target volume margins for brain metastases patients undergoing treatment with single and multi-fraction stereotactic radiotherapy on the Perfexion™ Gamma Knife unit, as observed on volumetric cone-beam computed tomography (CBCT) scans

CONTACTS AND LOCATIONS:
Overall Officials: David Shultz, M.D., Ph.D, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada